CLINICAL TRIAL: NCT00316524
Title: A Partially Randomized, Partially Double-blind, Placebo-controlled Phase II Non-inferiority Study to Evaluate Immunogenicity and Safety of One and Two Doses of MVA-BN® (IMVAMUNE™) Smallpox Vaccine in 18-55 Year Old Healthy Subjects
Brief Title: A Randomized, Double-blind, Placebo-controlled Study on Immunogenicity and Safety of MVA-BN (IMVAMUNE™) Smallpox Vaccine in Healthy Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bavarian Nordic (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: POX-MVA-005; DMID 05-0128; EudraCT No. 2005-001781-14
Record Dates: First submitted 2006-04-19; First posted 2006-04-21 (Estimated); Results first posted 2019-01-09 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-02

CONDITIONS: Smallpox
Keywords: Smallpox; Vaccination; Prevention
MeSH Terms: conditions — Smallpox | interventions — smallpox and monkeypox vaccine modified vaccinia ankara-bavarian nordic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- GP 1: two x 1x10E08 TCID, MVA-BN® s.c., vaccinia naive (Experimental): vaccinia naive subjects receiving two subcutanenous vaccinations with 0.5ml MVA-BN® IMVAMUNE (1x10E08 TCID)
  Interventions: Biological: MVA-BN® (IMVAMUNE)
- GP 2: 1x10E08 TCID, MVA-BN®, 1x Placebo, s.c., vaccinia naive (Experimental): vaccinica naive subjects receiving one vaccination with 0.5ml MVA-BN® IMVAMUNE(1x10E08 TCID), followed by one vaccination Placebo (0.5ml Tris Buffer)
  Interventions: Biological: MVA-BN® (IMVAMUNE); Biological: Placebo
- GP 3: two x Placebo, s.c., vaccinia naive (Placebo Comparator): vaccinia naive subjects, receiving two subcutaneous vaccinations with Placebo (0.5ml Tris Buffer).
  Interventions: Biological: Placebo
- GP 4: 1x10E08 TCID, MVA-BN®, s.c., vaccinia experienced (Experimental): vaccinia experienced subjects, receiving one subcutaneous vaccination with 0.5ml MVA-BN® IMVAMUNE (1x10E08 TCID).
  Interventions: Biological: MVA-BN® (IMVAMUNE)

INTERVENTIONS:
Biological: MVA-BN® (IMVAMUNE) — 1x 10E8_TCID50
  Arms: GP 1: two x 1x10E08 TCID, MVA-BN® s.c., vaccinia naive; GP 2: 1x10E08 TCID, MVA-BN®, 1x Placebo, s.c., vaccinia naive; GP 4: 1x10E08 TCID, MVA-BN®, s.c., vaccinia experienced
Biological: Placebo — Tris-Buffer
  Arms: GP 2: 1x10E08 TCID, MVA-BN®, 1x Placebo, s.c., vaccinia naive; GP 3: two x Placebo, s.c., vaccinia naive

SUMMARY:
The primary objective of this study is to evaluate the immune response after a single vaccination of pre-immune subjects compared to two vaccinations in naive subjects.

In addition the study further investigates the cardiac safety profile of MVA-BN® in a healthy population compared to placebo.

DETAILED DESCRIPTION:
The study consists of 4 groups, which receive either MVA-BN once, MVA-BN two times, MVA-BN followed by placebo, or two administrations of placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects between 18 and 55 years of age.
2. Women must have a negative serum pregnancy test at screening and a negative urine or serum pregnancy test within 24 hours prior to vaccination.
3. Women of childbearing potential must have used an acceptable method of contraception for 30 days prior to the first vaccination, must agree to use an acceptable method of contraception during the study, and must not become pregnant for at least 28 days after the last vaccination. A woman is considered of childbearing potential unless post-menopausal or surgically sterilized. (Acceptable contraception methods are restricted to abstinence, barrier contraceptives, intrauterine contraceptive devices or licensed hormonal products.)
4. Lab values without clinically significant findings
5. Electrocardiogram (ECG) without abnormal findings (e.g. any kind of atrioventricular or intraventricular conditions or blocks such as complete left or right bundle branch block, AV-node block, QTc or PR prolongation, premature atrial contractions or other atrial arrhythmia, sustained ventricular arrhythmia, 2 premature ventricular contractions (PVC) in a row, ST elevation consistent with ischemia).

Groups 1, 2 and 3 (All vaccinia-naïve subjects) additionally:

1. No history of known or suspected previous smallpox vaccination.
2. No detectable vaccinia scar.

Group 4 (All previously vaccinated subjects) additionally:

1. History of previous smallpox vaccination (documented and/or typical vaccinia scar).
2. Most recent smallpox vaccination ≥ 5 years.

Exclusion Criteria:

1. Uncontrolled serious infection i.e. not responding to antimicrobial therapy.
2. History of or active autoimmune disease. Persons with vitiligo or thyroid disease taking thyroid replacement are not excluded.
3. Known or suspected impairment of immunologic function including, but not limited to, clinically significant liver disease; diabetes mellitus; moderate to severe kidney impairment.
4. History of malignancy, other than squamous cell or basal cell skin cancer, unless there has been surgical excision that is considered to have achieved cure. Subjects with history of skin cancer at the vaccination site are excluded.
5. History of coronary heart disease, myocardial infarction, angina, congestive heart failure, cardiomyopathy, stroke or transient ischemic attack, uncontrolled high blood pressure, or any other heart condition under the care of a doctor.
6. History of an immediate family member (father, mother, brother, or sister) who died due to ischemic heart disease before age 50 years.
7. Ten percent or greater risk of developing a myocardial infarction or coronary death within the next 10 years using the National Cholesterol Education Program's risk assessment tool. (http://hin.nhlbi.nih.gov/atpiii/calculator.asp?usertype=prof) NOTE: This criterion applies only to volunteers 20 years of age and older.
8. History of anaphylaxis or severe allergic reaction.
9. Immune modulatory therapy.
10. History of any serious medical condition, which in the opinion of the investigator would compromise the safety of the subject.
11. History or clinical manifestation of clinically significant and severe hematological, renal, hepatic, pulmonary, central nervous, cardiovascular or gastrointestinal disorders.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 745 (Actual)
Dates: Start 2006-04 (Actual); Primary Completion 2007-02 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank von Sonnenburg, Prof, Principal Investigator — Section of International Medicine & Public Health, Department of Infectious Diseases and Tropical Medicine, Ludwig-Maximilians Unviersity Munich
Locations (1):
- Harrison Clinical Research GmbH, Munich, Bavaria, Germany

REFERENCES:
- [Result] Zitzmann-Roth EM, von Sonnenburg F, de la Motte S, Arndtz-Wiedemann N, von Krempelhuber A, Uebler N, Vollmar J, Virgin G, Chaplin P. Cardiac safety of Modified Vaccinia Ankara for vaccination against smallpox in a young, healthy study population. PLoS One. 2015 Apr 16;10(4):e0122653. doi: 10.1371/journal.pone.0122653. eCollection 2015. PMID 25879867
- [Derived] Ilchmann H, Samy N, Reichhardt D, Schmidt D, Powell JD, Meyer TPH, Silbernagl G, Nichols R, Weidenthaler H, De Moerlooze L, Chen L, Chaplin P. One- and Two-Dose Vaccinations With Modified Vaccinia Ankara-Bavarian Nordic Induce Durable B-Cell Memory Responses Comparable to Replicating Smallpox Vaccines. J Infect Dis. 2023 May 12;227(10):1203-1213. doi: 10.1093/infdis/jiac455. PMID 36408618

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: 2 x MVA-BN® s.c., Vaccinia Naive: vaccinia naive subjects receiving two subcutaneous vaccinations with 0.5mL MVA-BN® IMVAMUNE (1x10E08 TCID50)
- Group 2: 1x MVA-BN®, 1x Placebo, s.c., Vaccinia Naive: vaccinia naive subjects receiving one subcutaneous vaccination with 0.5mL MVA-BN® IMVAMUNE (1x10E08 TCID50), followed by one vaccination Placebo (0.5mL Tris Buffer)
- Group 3: Two x Placebo, s.c., Vaccinia Naive: vaccinia naive subjects receiving two subcutaneous vaccinations with Placebo (0.5mL Tris Buffer).
  Placebo: Tris-Buffer
- Group 4: 1x MVA-BN®, s.c., Vaccinia Experienced: vaccinia experienced subjects receiving one subcutaneous vaccination with 0.5ml MVA-BN® IMVAMUNE (1x10E08 TCID50).
Period: Overall Study
Arm/Group | Group 1: 2 x MVA-BN® s.c., Vaccinia Naive | Group 2: 1x MVA-BN®, 1x Placebo, s.c., Vaccinia Naive | Group 3: Two x Placebo, s.c., Vaccinia Naive | Group 4: 1x MVA-BN®, s.c., Vaccinia Experienced
Started (Vaccinated) | 183 | 181 | 181 | 200
Completed (Active Trial Phase) | 175 | 173 | 175 | 200
Not Completed | 8 | 8 | 6 | 0

BASELINE CHARACTERISTICS:
Population: Safety Dataset
Groups:
- Group 1: 2x MVA-BN® s.c., Vaccinia Naive: vaccinia naive subjects receiving two subcutaneous vaccinations with 0.5mL MVA-BN® IMVAMUNE (1x10E08 TCID50)
- Group 3: 2x Placebo, s.c., Vaccinia Naive: vaccinia naive subjects receiving two subcutaneous vaccinations with Placebo (0.5mL Tris Buffer)
  Placebo: Tris-Buffer
- Total: Total of all reporting groups
Arm/Group | Group 1: 2x MVA-BN® s.c., Vaccinia Naive | Group 2: 1x MVA-BN®, 1x Placebo, s.c., Vaccinia Naive | Group 3: 2x Placebo, s.c., Vaccinia Naive | Group 4: 1x MVA-BN®, s.c., Vaccinia Experienced | Total
Number analyzed (Participants) | 183 | 181 | 181 | 200 | 745
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.3 (4.98) | 25.4 (4.38) | 26.0 (5.1) | 41.5 (7.59) | 29.8 (9.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 112 | 107 | 115 | 431
  Male | 86 | 69 | 74 | 85 | 314
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnic group: Caucasian | 178 | 176 | 177 | 198 | 729
  Ethnic group: Asian | 1 | 2 | 1 | 0 | 4
  Ethnic group: Black | 0 | 1 | 0 | 1 | 2
  Ethnic group: Arabic | 2 | 1 | 1 | 0 | 4
  Ethnic group: Other | 2 | 1 | 2 | 1 | 6
Region of Enrollment [Number; unit: participants]
  Germany | 183 | 181 | 181 | 200 | 745

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Seroconversion by ELISA
Description: Seroconversion rate based on vaccinia-specific Enzyme-linked Immunosorbent Assay (ELISA). Seroconversion is defined as the appearance of antibody titers ≥ detection limit (50) for initially seronegative subjects, or a doubling or more of the antibody titer compared to Baseline titer for initially seropositive subjects. Percentages based on number of subjects with data available.
Time Frame: 2 weeks following the last vaccination (Week 6 for Groups 1-3, Week 2 for Group 4)
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Groups:
- GP 1: Two x 1x10E08 TCID, MVA-BN® s.c., Vaccinia Naive: vaccinia naive subjects receiving two subcutaneous vaccinations with 0.5ml MVA-BN® IMVAMUNE (1x10E08 TCID)
  MVA-BN® (IMVAMUNE): 1x 10E8_TCID50
- GP 2: 1x10E08 TCID, MVA-BN®, 1x Placebo, s.c., Vaccinia Naive: vaccinia naive subjects receiving one subcutaneous vaccination with 0.5ml MVA-BN® IMVAMUNE (1x10E08 TCID), followed by one subcutaneous vaccination Placebo (0.5ml Tris Buffer)
  MVA-BN® (IMVAMUNE): 1x 10E8_TCID50
  Placebo: Tris-Buffer
- GP 3: Two x Placebo, s.c., Vaccinia Naive: vaccinia naive subjects receiving two subcutaneous vaccinations with Placebo (0.5ml Tris Buffer)
  Placebo: Tris-Buffer
- GP 4: 1x10E08 TCID, MVA-BN®, s.c., Vaccinia Experienced: vaccinia experienced subjects receiving one subcutaneous vaccination with 0.5ml MVA-BN® IMVAMUNE (1x10E08 TCID)
  MVA-BN® (IMVAMUNE): 1x 10E8_TCID50
Arm/Group | GP 1: Two x 1x10E08 TCID, MVA-BN® s.c., Vaccinia Naive | GP 2: 1x10E08 TCID, MVA-BN®, 1x Placebo, s.c., Vaccinia Naive | GP 3: Two x Placebo, s.c., Vaccinia Naive | GP 4: 1x10E08 TCID, MVA-BN®, s.c., Vaccinia Experienced
Number analyzed (Participants) | 176 | 174 | 175 | 200
percentage of subjects | 98.9 [96.0 to 99.9] | 82.2 [75.7 to 87.6] | 3.4 [1.3 to 7.3] | 95.5 [91.6 to 97.9]
Statistical Analysis 1: Comparison: GP 1: Two x 1x10E08 TCID, MVA-BN® s.c., Vaccinia Naive vs GP 4: 1x10E08 TCID, MVA-BN®, s.c., Vaccinia Experienced; Test type: Non-Inferiority — The non-inferiority margin to show that Group 4 (vaccinia experienced subjects receiving a single vaccination) is non-inferior to Group 1 (vaccinia naive subjects receiving 2 vaccinations) in terms of seroconversion rate 2 weeks after the last vaccination was predefined as -5% for the difference in seroconversion rates; Difference in seroconversion rates (%) = -3.4, 97.5% CI 1-sided [lower limit -7.36]

2. Primary Outcome: Number of Participants With ECG Changes
Description: Occurrence of any specific or unspecific ECG change. Assessments at Screening (SCR), Visit 2 (Week 2) and Visit 4 (Week 6).
Time Frame: within 2 weeks after each vaccination
Population: Safety dataset
Measure: Number; unit: participants
Groups:
- Group 2: 1x MVA-BN®, 1x Placebo, s.c., Vaccinia Naive: vaccinia naive subjects receiving one subcutaneous vaccination with 0.5mL MVA-BN® IMVAMUNE (1x10E08 TCID50), followed by one subcutaneous vaccination Placebo (0.5mL Tris Buffer)
Arm/Group | Group 1: 2x MVA-BN® s.c., Vaccinia Naive | Group 2: 1x MVA-BN®, 1x Placebo, s.c., Vaccinia Naive | Group 3: 2x Placebo, s.c., Vaccinia Naive | Group 4: 1x MVA-BN®, s.c., Vaccinia Experienced
Number analyzed (Participants) | 183 | 181 | 181 | 200
participants
  SCR : Supraventricular arrhytmia | 0 | 0 | 0 | 0
  SCR : Ventricular arrhythmia | 0 | 0 | 0 | 0
  SCR : AV block (PQ time >0.20 sec) 1st degree | 0 | 0 | 1 | 1
  SCR : Right bundle branch block - incomplete | 10 | 18 | 4 | 1
  SCR : ST elevation | 5 | 1 | 4 | 1
  SCR : ST depression | 0 | 1 | 0 | 1
  SCR : T inversion - pathological | 42 | 54 | 50 | 48
  SCR : T inversion - other | 14 | 19 | 22 | 16
  SCR : Low voltage | 0 | 0 | 0 | 1
  SCR : Other non-specific changes | 23 | 23 | 26 | 5
  SCR : Bradycardia | 30 | 28 | 30 | 6
  SCR : Arrhythmia | 4 | 3 | 8 | 1
  SCR : Repolarisation | 3 | 3 | 3 | 0
  SCR : Q-Abnormalities | 1 | 1 | 0 | 4
  SCR : Tall T-waves | 0 | 0 | 0 | 0
  Week 2 : Supraventricular arrhytmia | 0 | 1 | 0 | 0
  Week 2 : Ventricular arrhythmia | 0 | 1 | 1 | 0
  Week 2 : AV block (PQ time >0.20 sec) 1st degree | 0 | 0 | 1 | 1
  Week 2 : Right bundle branch block - incomplete | 9 | 17 | 15 | 15
  Week 2 : ST elevation | 3 | 1 | 2 | 0
  Week 2 : ST depression | 0 | 1 | 1 | 1
  Week 2 : T inversion - pathological | 34 | 46 | 40 | 31
  Week 2 : T inversion - other | 11 | 9 | 10 | 7
  Week 2 : Low voltage | 0 | 0 | 0 | 0
  Week 2 : Other non-specific changes | 34 | 29 | 34 | 14
  Week 2 : Bradycardia | 31 | 25 | 33 | 6
  Week 2 : Arrhythmia | 4 | 4 | 2 | 5
  Week 2 : Repolarisation | 1 | 3 | 2 | 1
  Week 2 : Q-Abnormalities | 0 | 3 | 1 | 4
  Week 2 : Tall T-waves | 1 | 3 | 0 | 0
  Week 6 : Supraventricular arrhytmia | 1 | 1 | 0 | NA — Visit not applicable to Group 4 subjects
  Week 6 : Ventricular arrhythmia | 0 | 0 | 0 | NA — Visit not applicable to Group 4 subjects
  Week 6 : AV block (PQ time >0.20 sec) 1st degree | 2 | 0 | 1 | NA — Visit not applicable to Group 4 subjects
  Week 6 : Right bundle branch block - incomplete | 10 | 20 | 12 | NA — Visit not applicable to Group 4 subjects
  Week 6 : ST elevation | 1 | 3 | 1 | NA — Visit not applicable to Group 4 subjects
  Week 6 : ST depression | 1 | 0 | 0 | NA — Visit not applicable to Group 4 subjects
  Week 6 : T inversion - pathological | 28 | 37 | 39 | NA — Visit not applicable to Group 4 subjects
  Week 6 : T inversion - other | 3 | 5 | 4 | NA — Visit not applicable to Group 4 subjects
  Week 6 : Low voltage | 0 | 0 | 0 | NA — Visit not applicable to Group 4 subjects
  Week 6 : Other non-specific changes | 35 | 35 | 33 | NA — Visit not applicable to Group 4 subjects
  Week 6 : Bradycardia | 30 | 23 | 28 | NA — Visit not applicable to Group 4 subjects
  Week 6 : Arrhythmia | 4 | 4 | 2 | NA — Visit not applicable to Group 4 subjects
  Week 6 : Repolarisation | 2 | 3 | 7 | NA — Visit not applicable to Group 4 subjects
  Week 6 : Q-Abnormalities | 1 | 0 | 1 | NA — Visit not applicable to Group 4 subjects
  Week 6 : Tall T-waves | 1 | 1 | 2 | NA — Visit not applicable to Group 4 subjects

3. Primary Outcome: Number of Cardiac Adverse Events (Adverse Events of Special Interest [AESI])
Description: Occurrence and relationship of any other cardiac symptom at any time during the study
Time Frame: within 32 weeks
Population: Safety dataset
Measure: Number; unit: events
Arm/Group | Group 1: 2x MVA-BN® s.c., Vaccinia Naive | Group 2: 1x MVA-BN®, 1x Placebo, s.c., Vaccinia Naive | Group 3: 2x Placebo, s.c., Vaccinia Naive | Group 4: 1x MVA-BN®, s.c., Vaccinia Experienced
Number analyzed (Participants) | 183 | 181 | 181 | 200
events
  Sinus tachycardia : related | 0 | 0 | 0 | 0
  Sinus tachycardia : unrelated | 1 | 1 | 0 | 0
  Tachycardia : related | 0 | 1 | 0 | 1
  Tachycardia : unrelated | 1 | 0 | 0 | 1
  Palpitations : related | 0 | 1 | 0 | 2
  Palpitations : unrelated | 1 | 1 | 1 | 3
  Mild pericardial effusion : related | 0 | 0 | 0 | 0
  Mild pericardial effusion : unrelated | 0 | 0 | 0 | 1

4. Secondary Outcome: Percentage of Participants With Seroconversion by ELISA
Description: as for outcome 1
Time Frame: 4 weeks following the last vaccination (Week 8 for Groups 1-3, Week 4 for Group 4)
Population: Full Analysis Set (includes subjects with data available 4 weeks following the last vaccination)
Measure: Number; unit: percentage of subjects
Arm/Group | Group 1: 2x MVA-BN® s.c., Vaccinia Naive | Group 2: 1x MVA-BN®, 1x Placebo, s.c., Vaccinia Naive | Group 3: 2x Placebo, s.c., Vaccinia Naive | Group 4: 1x MVA-BN®, s.c., Vaccinia Experienced
Number analyzed (Participants) | 178 | 175 | 177 | 199
percentage of subjects | 98.9 | 72.0 | 2.8 | 93.0

5. Secondary Outcome: Percentage of Participants With Seroconversion by PRNT
Description: Seroconversion rate based on vaccinia-specific Plaque Reduction Neutralization Test (PRNT). Seroconversion is defined as the appearance of antibody titers ≥ detection limit (6) for initially seronegative subjects, or a doubling or more of the antibody titer compared to Baseline titer for initially seropositive subjects. Percentages based on number of subjects with data available.
Time Frame: 2 weeks following the last vaccination (Week 6 for Groups 1-3, Week 2 for Group 4)
Population: Full Analysis Set
Measure: Number; unit: percentage of subjects
Arm/Group | Group 1: 2x MVA-BN® s.c., Vaccinia Naive | Group 2: 1x MVA-BN®, 1x Placebo, s.c., Vaccinia Naive | Group 3: 2x Placebo, s.c., Vaccinia Naive | Group 4: 1x MVA-BN®, s.c., Vaccinia Experienced
Number analyzed (Participants) | 176 | 174 | 175 | 200
percentage of subjects | 89.2 | 56.3 | 0.0 | 78.5

6. Secondary Outcome: Percentage of Participants With Seroconversion by PRNT
Description: as for outcome 5
Time Frame: 4 weeks following the last vaccination (Week 8 for Groups 1-3, Week 4 for Group 4)
Population: Full Analysis Set (includes subjects with data available 4 weeks following the last vaccination)
Measure: Number; unit: percentage of subjects
Arm/Group | Group 1: 2x MVA-BN® s.c., Vaccinia Naive | Group 2: 1x MVA-BN®, 1x Placebo, s.c., Vaccinia Naive | Group 3: 2x Placebo, s.c., Vaccinia Naive | Group 4: 1x MVA-BN®, s.c., Vaccinia Experienced
Number analyzed (Participants) | 178 | 175 | 177 | 199
percentage of subjects | 86.0 | 47.4 | 0.0 | 69.8

7. Secondary Outcome: Number of Participants With Related Serious Adverse Events
Description: Number of participants with any serious adverse event possibly, probably or definitely related to the study vaccine at any time during the study
Time Frame: within 32 weeks
Population: Safety dataset
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: 2x MVA-BN® s.c., Vaccinia Naive | Group 2: 1x MVA-BN®, 1x Placebo, s.c., Vaccinia Naive | Group 3: 2x Placebo, s.c., Vaccinia Naive | Group 4: 1x MVA-BN®, s.c., Vaccinia Experienced
Number analyzed (Participants) | 183 | 181 | 181 | 200
Participants | 1 | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Solicited Local Adverse Events
Description: Number of participants with solicited local AEs (pain, erythema, swelling and induration) within 8 days after any vaccination (vaccinations for Groups 1-3: Days 0 and 28; Group 4: Day 0). Percentages based on subjects with at least one completed diary card.
Time Frame: within 8 days after any vaccination
Population: Safety dataset
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: 2x MVA-BN® s.c., Vaccinia Naive | Group 2: 1x MVA-BN®, 1x Placebo, s.c., Vaccinia Naive | Group 3: 2x Placebo, s.c., Vaccinia Naive | Group 4: 1x MVA-BN®, s.c., Vaccinia Experienced
Number analyzed (Participants) | 182 | 179 | 179 | 200
Participants
  Injection site pain | 166 | 155 | 37 | 167
  Injection site erythema | 166 | 146 | 39 | 169
  Injection site swelling | 149 | 103 | 10 | 149
  Injection site induration | 162 | 146 | 5 | 155

9. Secondary Outcome: Number of Participants With Solicited General Adverse Events
Description: Number of participants with solicited systemic/general AEs (body temperature increased, headache, myalgia, nausea, and fatigue) within 8 days after any vaccination (vaccinations for Groups 1-3: Days 0 and 28; Group 4: Day 0). Percentages based on subjects with at least one completed diary card.
Time Frame: within 8 days after any vaccination
Population: Safety dataset
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: 2x MVA-BN® s.c., Vaccinia Naive | Group 2: 1x MVA-BN®, 1x Placebo, s.c., Vaccinia Naive | Group 3: 2x Placebo, s.c., Vaccinia Naive | Group 4: 1x MVA-BN®, s.c., Vaccinia Experienced
Number analyzed (Participants) | 182 | 179 | 179 | 200
Participants
  Body temperature increased | 18 | 21 | 10 | 10
  Headache | 60 | 84 | 49 | 53
  Myalgia | 29 | 22 | 20 | 42
  Nausea | 17 | 22 | 13 | 18
  Fatigue | 68 | 59 | 55 | 78

10. Secondary Outcome: Number of Participants With Related Grade>=3 Adverse Events
Description: Number of participants with any Grade >=3 AE probably, possibly, or definitely related to the study vaccine within 4 weeks after any vaccination (vaccinations for Groups 1-3: Days 0 and 28; Group 4: Day 0). Pooled solicited (local and general) and unsolicited AEs.
Time Frame: within 4 weeks after any vaccination
Population: Safety dataset
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: 2x MVA-BN® s.c., Vaccinia Naive | Group 2: 1x MVA-BN®, 1x Placebo, s.c., Vaccinia Naive | Group 3: 2x Placebo, s.c., Vaccinia Naive | Group 4: 1x MVA-BN®, s.c., Vaccinia Experienced
Number analyzed (Participants) | 183 | 181 | 181 | 200
Participants | 10 | 5 | 5 | 15

11. Secondary Outcome: Number of Participants With Unsolicited Non-serious Adverse Events
Description: Number of participants with non-serious unsolicited AEs within 4 weeks after any vaccination (vaccinations for Groups 1-3: Days 0 and 28; Group 4: Day 0).
Time Frame: within 4 weeks after any vaccination
Population: Safety dataset
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: 2x MVA-BN® s.c., Vaccinia Naive | Group 2: 1x MVA-BN®, 1x Placebo, s.c., Vaccinia Naive | Group 3: 2x Placebo, s.c., Vaccinia Naive | Group 4: 1x MVA-BN®, s.c., Vaccinia Experienced
Number analyzed (Participants) | 183 | 181 | 181 | 200
Participants | 113 | 106 | 78 | 99

ADVERSE EVENTS:
Time Frame: 32 weeks
Arm/Group | GP 1: Two x 1x10E08 TCID, MVA-BN® s.c., Vaccinia Naive | GP 2: 1x10E08 TCID, MVA-BN®, 1x Placebo, s.c., Vaccinia Naive | GP 3: Two x Placebo, s.c., Vaccinia Naive | GP 4: 1x10E08 TCID, MVA-BN®, s.c., Vaccinia Experienced
All-Cause Mortality (participants affected / at risk) | 0/183 | 0/181 | 0/181 | 0/200
Serious Adverse Events (participants affected / at risk) | 3/183 | 3/181 | 5/181 | 1/200
Other Adverse Events (participants affected / at risk) | 91/183 | 88/181 | 54/181 | 73/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GP 1: Two x 1x10E08 TCID, MVA-BN® s.c., Vaccinia Naive (N=183) | GP 2: 1x10E08 TCID, MVA-BN®, 1x Placebo, s.c., Vaccinia Naive (N=181) | GP 3: Two x Placebo, s.c., Vaccinia Naive (N=181) | GP 4: 1x10E08 TCID, MVA-BN®, s.c., Vaccinia Experienced (N=200)
Sarcoidosis (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thyroid cyst (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mental disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thyroidectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GP 1: Two x 1x10E08 TCID, MVA-BN® s.c., Vaccinia Naive (N=183) | GP 2: 1x10E08 TCID, MVA-BN®, 1x Placebo, s.c., Vaccinia Naive (N=181) | GP 3: Two x Placebo, s.c., Vaccinia Naive (N=181) | GP 4: 1x10E08 TCID, MVA-BN®, s.c., Vaccinia Experienced (N=200)
Headache (Nervous system disorders) | 10 (11) | 16 (17) | 11 (11) | 6 (6)
Injection site pruritus (General disorders) | 43 (61) | 36 (37) | 4 (4) | 49 (49)
Injection site hematoma (General disorders) | 6 (6) | 9 (9) | 5 (5) | 4 (4)
Injection site warmth (General disorders) | 9 (10) | 5 (5) | 0 (0) | 8 (8)
Injection site discoloration (General disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (3) | 7 (7) | 2 (3) | 4 (4)
Lymphadenopaty (Blood and lymphatic system disorders) | 4 (5) | 4 (4) | 2 (2) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 4 (4) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 4 (4) | 3 (3) | 6 (6)
Bronchitis (Infections and infestations) | 3 (3) | 4 (4) | 2 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 42 (45) | 20 (20) | 26 (28) | 4 (4)
Rhinitis (Infections and infestations) | 3 (3) | 1 (1) | 4 (4) | 1 (1)
Tonsilitis (Infections and infestations) | 4 (4) | 5 (5) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 5 (5) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1) | 3 (3) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 9 (9) | 8 (9) | 4 (4)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes